CLINICAL TRIAL: NCT07366385
Title: Clinical Evaluation of the Validity of Occlusal Contact Area Measurement Using OccluSense With Versus Without Customizable Stabilizing Tray
Brief Title: OccluSense is Sensor Based System Used as a Digital Method for Occlusal Contact Analysis, and Basically Used Without Any Support of Its Sensor. Therefore the Aim of This Study is to Clinically Evaluate the Validity of a Customizable Stabilizing Tray to Support OccluSense Sensor in.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hala Zakaria, lecturer at prosthodontics department Faculty of Dentistry Cairo University, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 41-9-25
Record Dates: First submitted 2026-01-16; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Occlusal Analysis

STUDY DESIGN:
Intervention Model Description: 22 healthy dental students, all aged from 18-25 years, was recruited on a voluntary basis, from the faculty of dentistry Cairo University with the following inclusion criteria; intact arches, no missing teeth, and no TMD disorder. The exclusion criteria included students with less than 24 natural teeth, the presence of active orthodontic treatment, as it could interfere with the data acquisition process, the presence of fixed restorations, severe malocclusion, and those with orofacial pain.
  The digital occlusal analysis device used in this study is the OccluSense® (Bausch, Cologne, Germany). Participants were divided into two groups; for group (A) the occlusal contacts was recoded using the osscluSense with customized centering tray, for group (B) the osscluSense was used without the customizable centering tray.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- osscluSense with customized centering tray (Experimental): occlusal contacts was recoded using the osscluSense with customized centering tray
  Interventions: Device: osscluSense with customized centering tray

INTERVENTIONS:
Device: osscluSense with customized centering tray — A customizable centering tray is a thermoplastic or 3D-printed tray designed to hold the OccluSense sensor straight and centered between arches

SUMMARY:
Background: Occlusal contacts analysis is of prime importance in order to perform an effective prosthetic restoration. Quantitative methods for occlusal contact analysis involve using digital systems to measure and analyze occlusal contacts and forces with greater precision than traditional methods. One of these devices is the OccluSense which is sensor based system and basically used without any support of its sensor. Therefore the aim of this study is to clinically evaluate the validity of a customizable stabilizing tray to support the sensor of the OccluSense intraoral. A total of 22 healthy dental students, aged from 18-25 years, are recruited. Each participant will undergo two set of recordings; firstly by the OccluSense without centering tray then with the tray seated intraoral. Occlusal contacts were recorded under maximum bite force and Maximum Intercuspation Position (MIP).

ELIGIBILITY:
Inclusion Criteria:

- intact arches, no missing teeth, and no TMD disorder.

Exclusion Criteria:

* patients with less than 24 natural teeth, the presence of active orthodontic treatment, as it could interfere with the data acquisition process, the presence of fixed restorations, severe malocclusion, and those with orofacial pain.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2025-09-01 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-11-30 (Actual)

PRIMARY OUTCOMES:
total number of occlusal contacts recorded by the device | this study has unique characteristics. Each participant underwent two set of occlusal recordings with one week interval between the intervention and control toto minimize the risk of muscle fatigue. the outcomes were measured and analyzed instantly
total contact area and the Number of contact points | two visits with one week interval

CONTACTS AND LOCATIONS:
Locations (1):
- faculty of dentistry Cairo University, Cairo, Manyal, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Amin BK, Sedeeq HY. The Accuracy of Occlusal Analysis of Intraoral Scanner, Occlusense and Articulating Paper - A Comparative Study. Preprints [Internet]. 2025 Jul; Available from: https://doi.org/10.20944/preprints202507.1837.v1